CLINICAL TRIAL: NCT06302998
Title: Dexmedetomidine and Vasopressin (DEX-PRESSIN) for Reducing In-hospital Mortality in Septic Shock Patients: A Protocol for Randomized Controlled Trial (DecatSepsis-2)
Brief Title: Dexmedetomidine and Vasopressin in Septic Shock
Acronym: DecatSepsis-2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.111
Record Dates: First submitted 2024-02-25; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Standard of Care; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled superiority trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be nurses - not invovled in the study - will be unware about the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEX-PRESSIN (Experimental): This group will receive vasopressin as the first-line vasopressor. DEX will be started after hemodynamic stabilization if the heart rate is >90 beats per minute (bpm). NE infusion will be the second-line vasoactive drug.
  Interventions: Drug: DEX-PRESSIN
- Standard-of-care group (Active Comparator): This group will receive conventional treatment according to the Surviving Sepsis Campaign 2021 guidelines. This group will receive vasopressin as the second line after NE and will not receive dexmedetomidine.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: DEX-PRESSIN — This group will receive vasopressin as the first-line vasopressor. DEX will be started after hemodynamic stabilization if the heart rate is >90 beats per minute (bpm). NE infusion will be the second-line vasoactive drug.
  Arms: DEX-PRESSIN
Drug: Standard of Care — This group will receive conventional treatment according to the SSC 2021 guidelines. This group will receive vasopressin as the second line after NE and will not receive DEX.
  Other Names: Control group
  Arms: Standard-of-care group

SUMMARY:
Rudiger and Singer suggested strategies for refining adrenergic stress (decatecholaminization). They proposed the use of dexmedetomidine and vasopressin to reduce the catecholamine load during sepsis. The investigators will use vasopressin as the primary vasopressor and a heart rate-calibrated dexmedetomidine infusion in septic shock patients.

The investigators of the current study will use DEXPRESSIN in septic shock patients to investigate the effects of decatecholaminization on in-hospital mortality.

DETAILED DESCRIPTION:
The investigator will include 260 patients with septic shock. The study will compare the use of vasopressin as the first-line vasopressor in septic shock in addition to the dexmedetomidine infusion as in the DecatSepsis trial versus the standard of care. The standard of care is guided by the Surviving Sepsis campaign in 2021.

The main outcomes of the study are in-hospital mortality, norepinephrine equivalent dose, ICU scores, and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who develop septic shock in whom a vasopressor is initiated to maintain a mean arterial blood pressure (MAP) of ≥65 mmHg in the presence of sepsis (≥2 SIRS criteria plus suspicion or confirmation of infection).

Exclusion Criteria:

* Patient refusal or inability to obtain consent
* Failure of hemodynamic stabilization or hemoglobin <7 g/dL at the time of inclusion
* Severe cardiac dysfunction [i.e., ejection fraction (EF) <30%]
* History of heart block or patient on pacemaker
* Severe valvular heart disease
* Chronic liver disease (Child-Pugh classification C)
* Pregnancy
* Patients with traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
in-hospital mortality | throughout the hospitalization period on average 90 days.
  All-cause inhospital mortality as a binary outcome

SECONDARY OUTCOMES:
survival analysis | through out the hospitalization period or 28 days after inclusion if discharged from hosptia; before 28 days
  time to die using Kaplan Mier Curve
Norepinephrine Equivalent Dose (NED) | over the first three days after enrolment or death
  mean NED over the first three days after enrolment or death, whichever comes first; the NED of epinephrine will be estimated as a 1:1 ratio
Duration of vasopressor infusion in survivors | through out the hospitalization period or 28 days after inclusion if discharged from hosptial before 28 days
  Duration in hours from the start of the vasopressor (NE or vasopressin) infusion till the time of discontinuation.
Initiation of invasive mechanical ventilation (IMV) | through out the hospitalization period or 28 days after inclusion if discharged from hosptial before 28 days
  incidence of IMV
Duration of IMV | through out the hospitalization period or 28 days after inclusion if discharged from hosptial before 28 days
  duratioin in hours
Early acute kidney injury (AKI) | within 48 hours
  AKI according to the KDIGO guidelines 2012
Late acute kidney injury (AKI) | between 48 hours and 7 days
  AKI according to the KDIGO guidelines 2012
Acute Physiology and Chronic Health Evaluation (APACHE-II) | on the 3rd day after enrollment
  As a score on MedCalc
Simplified Acute Physiology Score (SAPS) II score | on the 3rd day after enrollment
  As a score on MedCalc
ICU length of stay | during hospitalization period on average 90 days
  duration in days in survivors
Hospital length of stay | during hospitlaization period on average 90 days
  duration in days in survivors

CONTACTS AND LOCATIONS:
Overall Officials: Moataz M Emara, Principal Investigator — Mansoura University Hospital

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual patients' data will be available with the prinicpal investigator on reasonable request after approval by the local IRB.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within 5 years after the study
Access Criteria: Undecided